CLINICAL TRIAL: NCT04073875
Title: 18F-GP1 Positron Emission Tomography-computed Tomography to Detect Bioprosthetic Aortic Valve Thrombosis; the Biothrombus Study.
Brief Title: 18F-GP1 PET-CT to Detect Bioprosthetic Aortic Valve Thrombosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Life Molecular Imaging SA (Industry); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: E181981
Record Dates: First submitted 2019-08-22; First posted 2019-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Thrombosis Cardiac; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bioprosthetic aortic valve: Single 18F-GP1 PET-CT
  Interventions: Diagnostic Test: 18F-GP1
- Bioprosthetic aortic valve thrombus - repeat imaging: 18F-GP1 PET-CT at baseline and 3 months
  Interventions: Diagnostic Test: 18F-GP1

INTERVENTIONS:
Diagnostic Test: 18F-GP1 — 18F-GP1 PET-CT scan

SUMMARY:
18F-GP1 binds with high affinity to the glycoprotein IIb/IIIa receptors on activated platelets. 18F-GP1 PET-CT has recently demonstrated favourable safety, pharmacokinetic, biodistribution and diagnostic performance for the in vivo identification of venous and arterial thrombemboli.

DETAILED DESCRIPTION:
Aortic stenosis is the most common reason for valvular interventions in the developed world, with rates projected to increase as the population ages. Aortic valve replacement remains the only recognised treatment available. Bioprostheses are far more common than mechanical prostheses, particularly with increasing rates of transcatheter heart valve use.

Bioprothetic valves are less durable than mechanical valves and are subject to deterioration which may lead to clinical heart failure and the need for re-intervention. Long-term results with surgical bioprostheses are well reported, with valve deterioration rates of less than 15% at 10 years. These data, however, rely on re-operation rather than echocardiographic measures, suggesting that the true incidence of structural valve deterioration is underestimated.

Valve thrombosis is increasingly recognised as a potential contributor to leaflet degeneration and has been detected in participants undergoing both surgical aortic valve replacement and transcatheter aortic valve implantation. The role of valve thrombosis as an early trigger for calcification and subsequent valve degeneration has not been addressed. The true incidence of valve thrombosis and its impact on clinical outcomes is unknown due to the lack of a sufficiently sensitive non-invasive imaging modality to detect early subclinical thrombosis. Current observational data suggests rates of 12 to 40%, based on computed tomography findings. There is a clinical need for a more sensitive non-invasive method of detecting valve thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* >1 month post-surgical or transcatheter aortic valve replacement

Exclusion Criteria:

* Inability to give informed consent
* Pregnancy or breastfeeding
* Contraindications to iodinated contrast
* Contraindications to anticoagulation
* Use of anticoagulants during the post-operative period prior to screening
* Extreme claustrophobia
* Chronic kidney disease (with estimated glomerular filtration rate <30 mL/min/1.73m2)
* Metastatic malignancy
* Inability to tolerate the supine position

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >1 month post-bioprosthetic aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Prevalence of 18F-GP1 PET-CT bioprosthetic aortic valve uptake | 2 years
  Prevalence of 18F-GP1 PET-CT bioprosthetic aortic valve uptake as measured by standardised uptake values.
Intensity of 18F-GP1 PET-CT activity in bioprosthetic aortic valve thrombus | 2 years
  Intensity of 18F-GP1 PET-CT activity in bioprosthetic aortic valve thrombus compared to blood pool as measured by standardised uptake values.

SECONDARY OUTCOMES:
18F-GP1 PET-CT bioprosthetic aortic valve uptake in patients with thrombus. | 2 years
  18F-GP1 PET-CT bioprosthetic aortic valve uptake after 3 months in patients with evidence of thrombus at baseline as measured by standardised uptake values.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohrke J, Siebeneicher H, Berger M, Reinhardt M, Berndt M, Mueller A, Zerna M, Koglin N, Oden F, Bauser M, Friebe M, Dinkelborg LM, Huetter J, Stephens AW. 18F-GP1, a Novel PET Tracer Designed for High-Sensitivity, Low-Background Detection of Thrombi. J Nucl Med. 2017 Jul;58(7):1094-1099. doi: 10.2967/jnumed.116.188896. Epub 2017 Mar 16. PMID 28302764
- [Background] Kim C, Lee JS, Han Y, Chae SY, Jin S, Sung C, Son HJ, Oh SJ, Lee SJ, Oh JS, Cho YP, Kwon TW, Lee DH, Jang S, Kim B, Koglin N, Berndt M, Stephens AW, Moon DH. Glycoprotein IIb/IIIa receptor imaging with 18F-GP1 positron emission tomography for acute venous thromboembolism: an open-label, non-randomized, first-in-human phase 1 study. J Nucl Med. 2018 Jun 29;60(2):244-9. doi: 10.2967/jnumed.118.212084. Online ahead of print. PMID 29959214
- [Background] Chae SY, Kwon TW, Jin S, Kwon SU, Sung C, Oh SJ, Lee SJ, Oh JS, Han Y, Cho YP, Lee N, Kim JY, Koglin N, Berndt M, Stephens AW, Moon DH. A phase 1, first-in-human study of 18F-GP1 positron emission tomography for imaging acute arterial thrombosis. EJNMMI Res. 2019 Jan 7;9(1):3. doi: 10.1186/s13550-018-0471-8. PMID 30617563
- [Background] Lee N, Oh I, Chae SY, Jin S, Oh SJ, Lee SJ, Koglin N, Berndt M, Stephens AW, Oh JS, Moon DH. Radiation dosimetry of [18F]GP1 for imaging activated glycoprotein IIb/IIIa receptors with positron emission tomography in patients with acute thromboembolism. Nucl Med Biol. 2019 May-Jun;72-73:45-48. doi: 10.1016/j.nucmedbio.2019.07.003. Epub 2019 Jul 10. PMID 31330411
- [Background] Durko AP, Osnabrugge RL, Van Mieghem NM, Milojevic M, Mylotte D, Nkomo VT, Pieter Kappetein A. Annual number of candidates for transcatheter aortic valve implantation per country: current estimates and future projections. Eur Heart J. 2018 Jul 21;39(28):2635-2642. doi: 10.1093/eurheartj/ehy107. PMID 29546396
- [Background] Johnston DR, Soltesz EG, Vakil N, Rajeswaran J, Roselli EE, Sabik JF 3rd, Smedira NG, Svensson LG, Lytle BW, Blackstone EH. Long-term durability of bioprosthetic aortic valves: implications from 12,569 implants. Ann Thorac Surg. 2015 Apr;99(4):1239-47. doi: 10.1016/j.athoracsur.2014.10.070. Epub 2015 Feb 4. PMID 25662439
- [Background] Rodriguez-Gabella T, Voisine P, Puri R, Pibarot P, Rodes-Cabau J. Aortic Bioprosthetic Valve Durability: Incidence, Mechanisms, Predictors, and Management of Surgical and Transcatheter Valve Degeneration. J Am Coll Cardiol. 2017 Aug 22;70(8):1013-1028. doi: 10.1016/j.jacc.2017.07.715. PMID 28818190
- [Background] Chakravarty T, Sondergaard L, Friedman J, De Backer O, Berman D, Kofoed KF, Jilaihawi H, Shiota T, Abramowitz Y, Jorgensen TH, Rami T, Israr S, Fontana G, de Knegt M, Fuchs A, Lyden P, Trento A, Bhatt DL, Leon MB, Makkar RR; RESOLVE; SAVORY Investigators. Subclinical leaflet thrombosis in surgical and transcatheter bioprosthetic aortic valves: an observational study. Lancet. 2017 Jun 17;389(10087):2383-2392. doi: 10.1016/S0140-6736(17)30757-2. Epub 2017 Mar 19. PMID 28330690
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Derived] Bing R, Deutsch MA, Sellers SL, Corral CA, Andrews JPM, van Beek EJR, Bleiziffer S, Burchert W, Clark T, Dey D, Friedrichs K, Gummert JF, Koglin N, Leipsic JA, Lindner O, MacAskill MG, Milting H, Pessotto R, Preuss R, Raftis JB, Rudolph TK, Rudolph V, Slomka P, Stephens AW, Tavares A, Tzolos E, Weir N, White AC, Williams MC, Zabel R, Dweck MR, Hugenberg V, Newby DE. 18F-GP1 Positron Emission Tomography and Bioprosthetic Aortic Valve Thrombus. JACC Cardiovasc Imaging. 2022 Jun;15(6):1107-1120. doi: 10.1016/j.jcmg.2021.11.015. Epub 2022 Jan 12. PMID 35033495